CLINICAL TRIAL: NCT00605176
Title: A Phase 3, Randomized, Double-blinded, Placebo-controlled, Multicenter, Efficacy and Safety Study of Four Weeks of Treatment With Imiquimod Creams for Actinic Keratoses
Brief Title: Safety and Effectiveness Study of Imiquimod Creams for Treatment of Actinic Keratoses (AKs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Vice President, Product Development, Clinical, Graceway Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW01-0702 / 0704
Record Dates: First submitted 2008-01-16; First posted 2008-01-30 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Actinic Keratoses
Keywords: Actinic keratosis; Skin disease
MeSH Terms: conditions — Keratosis, Actinic; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3.75% imiquimod cream (Active Comparator)
  Interventions: Drug: imiquimod cream
- 2.5% imiquimod cream (Active Comparator)
  Interventions: Drug: imiquimod cream
- Placebo cream (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: imiquimod cream — cream, 250 mg/packet, up to 2 packets applied daily for 2 treatment cycles. The first treatment cycle consisted of 2 weeks of daily treatment followed by 2 weeks of no treatment, and the second treatment cycle consisted of an additional 2 weeks of daily treatment followed by 8 weeks of no treatment.
  Arms: 3.75% imiquimod cream
Drug: imiquimod cream — cream, 250 mg/packet, up to 2 packets applied daily for 2 treatment cycles. The first treatment cycle consisted of 2 weeks of daily treatment followed by 2 weeks of no treatment, and the second treatment cycle consisted of an additional 2 weeks of daily treatment followed by 8 weeks of no treatment.
  Arms: 2.5% imiquimod cream
Drug: Placebo — cream, 250 mg/packet, up to 2 packets applied daily for 2 treatment cycles. The first treatment cycle consisted of 2 weeks of daily treatment followed by 2 weeks of no treatment, and the second treatment cycle consisted of an additional 2 weeks of daily treatment followed by 8 weeks of no treatment.
  Arms: Placebo cream

SUMMARY:
The purpose of this study is to determine whether imiquimod creams are effective in treating Actinic Keratoses when applied to the face or balding scalp.

Actinic keratosis (AK) is a skin condition that shows up on skin routinely exposed to the sun, such as the face, scalp, shoulders, chest, back, arms, and hands. The active ingredient contained in the study cream for this study is the same as that of the approved product Aldara, which has been shown to be safe and effective for the treatment of AKs.

DETAILED DESCRIPTION:
This was a randomized, double-blind, multicenter, placebo-controlled study that compared the efficacy and safety of 2.5% imiquimod cream and 3.75% imiquimod cream with that of placebo in the treatment of typical visible or palpable AKs of the face or balding scalp. Subjects were scheduled for a total of 9 visits (1 prestudy screening visit and 8 on-study visits). Subjects determined to be eligible during the screening phase were randomized in a 1:1:1 ratio to 2.5% imiquimod cream, 3.75% imiquimod cream, or placebo cream. The creams were applied daily for 2 treatment cycles. The first treatment cycle consisted of 2 weeks of daily treatment followed by 2 weeks of no treatment, and the second treatment cycle consisted of an additional 2 weeks of daily treatment followed by 8 weeks of no treatment. The investigator selected the treatment area for the study (either the entire face or the entire balding scalp, but not both). Subjects applied a thin layer of cream to the treatment area (up to 2 packets, or 500 mg of product, per application), avoiding the periocular areas, lips, and nares. Study medication was applied prior to normal sleeping hours and removed approximately 8 hours later with mild soap and water. Ears were excluded from both assessment and treatment. Rest periods from daily treatment were instituted by the investigator as needed to manage local skin reactions (LSRs) or application site reactions, with resumption of treatment upon adequate resolution as determined by the investigator.

The duration of each subject's study participation was approximately 18 weeks, including a 4-week maximum screening period and a 14-week study period.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Have 5 to 20 AKs on the face or balding scalp
* Negative urine pregnancy test (for women who are able to become pregnant)
* Willing to make frequent visits to the study center during treatment and follow-up periods.

Exclusion Criteria:

* Women who are pregnant, lactating or planning to become pregnant during the study.
* Have had a medical event within 90 days of the first visit (such as; stroke, heart attack).
* Have any skin condition in the treatment area that may be made worse by treatment with imiquimod (e.g., rosacea, psoriasis, atopic dermatitis, eczema).
* Have received specific treatments/medications in the treatment area(s) within the designated time period prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon F Levy, MD, Study Director — Graceway Pharmaceuticals
Locations (26):
- United States (26):
  - Fremont, California
  - Los Angeles, California
  - Riverside, California
  - San Diego, California
  - Vallejo, California
  - Miami, Florida
  - Newnan, Georgia
  - Boise, Idaho
  - Springfield, Illinois
  - Dubuque, Iowa
  - Olathe, Kansas
  - Wichita, Kansas
  - Marrero, Louisiana
  - Henderson, Nevada
  - Rochester, New York
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Lynchburg, Virginia

REFERENCES:
- [Result] Swanson N, Abramovits W, Berman B, Kulp J, Rigel DS, Levy S. Imiquimod 2.5% and 3.75% for the treatment of actinic keratoses: results of two placebo-controlled studies of daily application to the face and balding scalp for two 2-week cycles. J Am Acad Dermatol. 2010 Apr;62(4):582-90. doi: 10.1016/j.jaad.2009.07.004. Epub 2010 Feb 4. PMID 20133013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on January 15, 2008 all subjects were randomized by March 17, 2008. The studies were performed at 26 investigational centers in the United States.
Pre-assignment Details: Subjects were screened and had to meet eligibility requirements for randomization. The most frequent reason for screen failure (104 of screen failures) was that the subject did not have between 5 and 20 visible or palpable Actinic Keratosis (AK) lesions on either the face or the balding scalp.
Groups:
- 3.75% Imiquimod Cream; 2.5% Imiquimod Cream; Placebo Cream: 250 mg/packet, up to 2 packets applied daily for 2 treatment cycles. The first treatment cycle consisted of 2 weeks of daily treatment followed by 2 weeks of no treatment, and the second treatment cycle consisted of an additional 2 weeks of daily treatment followed by 8 weeks of no treatment.
Period: Overall Study
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream
Started | 160 | 160 | 159
Completed | 149 | 154 | 150
Not Completed | 11 | 6 | 9
Not completed — Adverse Event | 2 | 1 | 3
Not completed — Withdrawal by Subject | 4 | 2 | 4
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Non-complicance with study procedures | 1 | 0 | 0
Not completed — Use of concomitant therapy | 1 | 0 | 1
Not completed — Other (not due to AE) | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream | Total
Number analyzed (Participants) | 160 | 160 | 159 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 82 | 88 | 90 | 260
  >=65 years | 78 | 72 | 69 | 219
Age Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.6) | 64.3 (10.5) | 64.3 (8.9) | 64.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 33 | 29 | 90
  Male | 132 | 127 | 130 | 389
Region of Enrollment [Number; unit: participants]
  United States | 160 | 160 | 159 | 479

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Clearance of AK Lesions
Description: Subject status with respect to complete clearance of AK lesions at End of Study (EOS), ie, the Week 14 visit. Complete clearance was defined as the absence of clinically visible or palpable AK lesions in the treatment area. All lesions within the identified treatment area were included in the count, even if the lesion was a new lesion or 'subclinical' lesion that had not been identified at Baseline.
Time Frame: End of Study the Week 14 visit
Population: Efficacy analyses were conducted on the intent-to-treat (ITT) population. For the primary efficacy variable, imputations were made for missing data points using last observation carried forward (LOCF, primary analysis), taking all missed observations as failure (sensitivity analysis), and using observed cases only (supportive analysis).
Measure: Number; unit: participants
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream
Number analyzed (Participants) | 160 | 160 | 159
participants | 57 | 49 | 10

2. Secondary Outcome: Number of Participants With Partial Clearance of AK Lesions
Description: Subject status with respect to partial clearance of AK lesions at end of study (EOS), defined as at least a 75% reduction in the number of AK lesions in the treatment area compared with Baseline.
Time Frame: End of Study the Week 14 visit
Population: Efficacy analyses were conducted on the intent-to-treat (ITT) population. Imputations were made for missing data points using last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream
Number analyzed (Participants) | 160 | 160 | 159
participants | 95 | 77 | 36

3. Secondary Outcome: Percent Change From Baseline in AK Lesion Count
Description: Percent change from Baseline to end of study (EOS) in investigator counts of AK lesions.
Time Frame: From baseline to End of Study the Week 14 visit
Population: Intent to treat (ITT) Last Observation Carried Forward (LOCF)
Measure: Median (Full Range); unit: percent change
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream
Number analyzed (Participants) | 160 | 160 | 159
percent change | -81.8 [-100.0 to 188.9] | -71.8 [-100.0 to 90.0] | -25.0 [-100.0 to 300.0]

4. Secondary Outcome: Local Skin Reactions
Description: Six local skin reaction (LSR) signs were predefined and were assessed for presence and intensity at each study visit. These included: Erythema, Edema, Weeping/Exudate, Flaking/Scaling/Dryness, Scabbing/Crusting and Erosion/Ulceration. The LSRs were scored as 0=none, 1=mild, 2=moderate, 3=severe. Mean scores were summated over time (14 weeks) to yield a mean LSR AUC (area under the curve)
Time Frame: At all visits - from Baseline to End of study (Week 14)
Population: All participants were evaluated for local skin reactions (LSR) at every visit. Summary of LSR - area under the curve (AUC) of sum of LSR Scores (days). ITT population. The time period for the AUC extends to 8 weeks after the end of treatment (Week 14). Only subjects who received treatment in both treatment cycles are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale * days
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream
Number analyzed (Participants) | 148 | 158 | 153
units on a scale * days | 272.0 (123.0) | 242.5 (126.2) | 139.8 (104.1)

ADVERSE EVENTS:
Time Frame: From study screening through the last study visit. Day 1 (first study visit) through the end of study (Week 14 visit)
Description: Subjects were queried indirectly regarding AEs during each study visit.
Arm/Group | 3.75% Imiquimod Cream | 2.5% Imiquimod Cream | Placebo Cream
Serious Adverse Events (participants affected / at risk) | 5/160 | 5/160 | 2/159
Other Adverse Events (participants affected / at risk) | 14/160 | 7/160 | 13/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75% Imiquimod Cream (N=160) | 2.5% Imiquimod Cream (N=160) | Placebo Cream (N=159)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Small intestine obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75% Imiquimod Cream (N=160) | 2.5% Imiquimod Cream (N=160) | Placebo Cream (N=159)
Headache (Nervous system disorders) | 10 (10) | 3 (3) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No